CLINICAL TRIAL: NCT02389426
Title: Evaluation of Cerebrovascular Hemodynamics With Transcranial Doppler and Near-infrared Spectroscopy in Patients With Multiple Sclerosis
Brief Title: Transcranial Doppler in Multiple Sclerosis
Acronym: TRADOMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: B.U.N. 1432101422450
Record Dates: First submitted 2015-02-09; First posted 2015-03-17 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Cerebral hemodynamics; Cerebral hypoperfusion; Cerebral circulation
MeSH Terms: conditions — Multiple Sclerosis | interventions — Ultrasonography, Doppler, Transcranial; Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with Multiple Sclerosis (Experimental): One examination with TCD baseline and with NIRS baseline, and a second examination with TCD after bosentan administration and with NIRS after bosentan administration will be performed; The examination will be repeated only in the patients with MS (i.e. not in control subjects) 4 h after the oral intake of one tablet 62.5 mg bosentan (Tracleer®) (when peak plasma concentrations are expected).
  Interventions: Device: TCD baseline; Device: TCD after bosentan administration; Device: NIRS baseline; Device: NIRS after bosentan administration
- Healthy controls (Experimental): Only one examination with TCD baseline and NIRS baseline will be performed, without administration of bosentan.
  Interventions: Device: TCD baseline; Device: NIRS baseline

INTERVENTIONS:
Device: TCD baseline — Measurement of cerebral circulation parameters with transcranial doppler baseline.
  This examination will be performed in patients with multiple sclerosis and in healthy controls.
  Other Names: Transcranial doppler
Device: TCD after bosentan administration — Measurement of cerebral circulation parameters with transcranial doppler after administration of one tablet tracleer (Bosentan) 62,5 mg per oral.
  This examination will only be performed in patients with multiple sclerosis.
  Other Names: Transcranial doppler; Tracleer; Endothelin-1 receptor antagonist
  Arms: Patients with Multiple Sclerosis
Device: NIRS baseline — Measurement of frontal lobe oxygen saturation with near-infrared spectroscopy baseline.
  This examination will be performed in patients with multiple sclerosis and in healthy controls.
  Other Names: Near-infrared spectroscopy; ForeSight
Device: NIRS after bosentan administration — Measurement of frontal lobe oxygen saturation with near-infrared spectroscopy after administration of one tablet tracleer (Bosentan) 62,5 mg per oral.
  This examination will only be performed in patients with multiple sclerosis.
  Other Names: Near-infrared Spectroscopy; Endothelin-1 receptor antagonist; Tracleer
  Arms: Patients with Multiple Sclerosis

SUMMARY:
The aim of this study is to investigate the potential of Transcranial doppler (TCD) and Near-Infrared Spectroscopy (NIRS), more simple and non-invasive bedside methods than magnetic resonance imaging (MRI), to evaluate changes in the cerebral circulation between patients with MS and control subjects.

DETAILED DESCRIPTION:
MS is a poorly understood chronic disease of the central nervous system characterized by focal inflammatory demyelinating lesions and diffuse axonal degeneration. Recent magnetic resonance imaging (MRI) studies demonstrated a widespread decrease in cerebral perfusion - expressed as cerebral blood flow (CBF) - throughout the normal-appearing white matter of patients with MS, which seems not just to be secondary to axonal degeneration with reduced metabolic demands, but in contrast may actively contribute to MS pathology.

Reduced CBF in MS is mediated by elevated levels of the potent vasoconstrictive agent endothelin-1 (ET-1), likely released in the cerebral circulation by reactive astrocytes, and can reversed with administration of the ET-1 antagonist bosentan.

Phase-contrast MRI recently demonstrated reduced cervical arterial blood flow velocities to the brain in patients MS as compared to control subjects. The aim of this study is to investigate the potential of TCD and NIRS, more simple and non-invasive bedside method, to evaluate changes in the cerebral circulation between patients with MS and control subjects.

A baseline TCD examination will be performed in each subject (MS patients and controls) over the temporal bone window on both sides. Middle cerebral artery wave forms will be identified at a depth range of 40-60 mm and a stable forward waveform with good intensity will be selected. TCD probes (2 MHz) will be mounted by a head frame to ensure a constant angle of insonation throughout the procedure. Mean, peak-systolic and end-diastolic blood flow velocities can be directly recorded from the machine. Blood pressure (BP) and heart rate will be measured with a finger plethysmograph. The cuff will be applied to the middle finger of the left hand, first placed at the heart level to calibrate the system, afterwards the hand is placed next to the subject in rest. Near-infrared spectroscopy will be performed to measure cerebral frontal lobe oxygen saturation. NIRS is performed with two large sensors, attached on patient's forehead bilaterally. In bright environments, a light-blocker to cover the sensors will be used to reduce interference from ambient light. Continuously NIRS recording with a 2s interval refreshment. Measurements will be done in upright and supine positions. The expected duration of the entire TCD protocol is 30 minutes.

The TCD examination will be repeated only in the patients with MS (i.e. not in control subjects) 4 h after the oral intake of 62.5 mg bosentan (Tracleer®) (when peak plasma concentrations are expected). This is a purely academic study and Bosentan will be purchased through the hospital pharmacy. The most common side effect of daily treatment with bosentan is hepatotoxicity. Adverse reactions to one single dose are very unlikely. The primary aim is to investigate the potential of TCD to evaluate changes in the cerebral circulation between patients with MS and controls. Bosentan is not the object of investigation in this study but can be considered as a 'Non Investigational Medicinal Product' (N.I.M.P.). Patients with MS will receive the product to increase CBF, an effect which has already been demonstrated in an earlier perfusion-weighted MRI study.

Fifteen patients with relapsing-remitting or progressive MS and 15 healthy controls, matched for sex and age, will be included in this study. Sample size calculation is based on the number of inclusion in previous studies regarding cerebral hemodynamic parameters in MS (mostly between 10 and 30).

The statistical analyses will be conducted with Statistical Package for the Social Sciences (SPSS) software. Mann Whitney U or Wilcoxon signed rank tests will be used where appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of relapsing-remitting, primary progressive of secondary progressive MS, according to the 2010 revised McDonald criteria.
* Written informed consent must be obtained.

Exclusion Criteria:

* MS patients with a known contra-indication for bosentan: liver dysfunction, use of cyclosporine A, allergy.
* Pregnancy
* No evidence of MS relapse within the 3 months prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-12; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Detection of hemodynamic differences between MS patients and Healthy controls with TCD baseline. | a 10 minute recording with TCD baseline
  Evaluation of cerebral circulation parameters altogether with measured blood pressure and heart rate values.

SECONDARY OUTCOMES:
Hemodynamic changes in MS patients detected with TCD after administration of Bosentan | baseline and 4 hours after administration of bosentan a 10 minute recording with TCD
  Evaluation of cerebral circulation parameters altogether with measured blood pressure and heart rate values in MS patients, compared before and after administration of bosentan.
Detection of frontal lobe oxygen saturation differences between patients with multiple sclerosis and healthy controls with near-infrared spectroscopy. | a 10 minute recording with NIRS baseline
  Analysis of oxygen saturation measurements of the left and right frontal cerebral lobe.
Frontal lobe oxygen saturation changes in MS patients detected with NIRS after administration of Bosentan | baseline and 4 hours after administration of bosentan a 10 minute recording with NIRS
  Analysis of oxygen saturation measurements of the left and right frontal cerebral lobe in MS patients, compared before and after administration of bosentan.

CONTACTS AND LOCATIONS:
Overall Officials: Ilse AS Peeters, Student, Principal Investigator — Department of Neurology, Universitair Ziekenhuis (UZ) Brussel, Brussels. Belgium Center for Neurosciences, Vrije Universiteit Brussel, Brussels, Belgium; Miguel D'haeseleer, MD, PhD, Study Chair — Department of Neurology, Universitair Ziekenhuis (UZ) Brussel, Brussels. Belgium Center for Neurosciences, Vrije Universiteit Brussel, Brussels, Belgium; Jacques De Keyser, MD, PhD, Study Director — Department of Neurology, Universitair Ziekenhuis (UZ) Brussel, Brussels. Belgium Center for Neurosciences, Vrije Universiteit Brussel, Brussels, Belgium
Locations (1):
- Department of Neurology, Universitair Ziekenhuis (UZ) Brussel. Center for Neurosciences, Vrije Universiteit Brussel, Jette, Vlaams-Brabant, Belgium

REFERENCES:
- [Background] Law M, Saindane AM, Ge Y, Babb JS, Johnson G, Mannon LJ, Herbert J, Grossman RI. Microvascular abnormality in relapsing-remitting multiple sclerosis: perfusion MR imaging findings in normal-appearing white matter. Radiology. 2004 Jun;231(3):645-52. doi: 10.1148/radiol.2313030996. PMID 15163806
- [Background] Adhya S, Johnson G, Herbert J, Jaggi H, Babb JS, Grossman RI, Inglese M. Pattern of hemodynamic impairment in multiple sclerosis: dynamic susceptibility contrast perfusion MR imaging at 3.0 T. Neuroimage. 2006 Dec;33(4):1029-35. doi: 10.1016/j.neuroimage.2006.08.008. Epub 2006 Sep 22. PMID 16996280
- [Background] Varga AW, Johnson G, Babb JS, Herbert J, Grossman RI, Inglese M. White matter hemodynamic abnormalities precede sub-cortical gray matter changes in multiple sclerosis. J Neurol Sci. 2009 Jul 15;282(1-2):28-33. doi: 10.1016/j.jns.2008.12.036. Epub 2009 Jan 31. PMID 19181347
- [Background] Saindane AM, Law M, Ge Y, Johnson G, Babb JS, Grossman RI. Correlation of diffusion tensor and dynamic perfusion MR imaging metrics in normal-appearing corpus callosum: support for primary hypoperfusion in multiple sclerosis. AJNR Am J Neuroradiol. 2007 Apr;28(4):767-72. PMID 17416836
- [Background] D'haeseleer M, Beelen R, Fierens Y, Cambron M, Vanbinst AM, Verborgh C, Demey J, De Keyser J. Cerebral hypoperfusion in multiple sclerosis is reversible and mediated by endothelin-1. Proc Natl Acad Sci U S A. 2013 Apr 2;110(14):5654-8. doi: 10.1073/pnas.1222560110. Epub 2013 Mar 18. PMID 23509249
- [Background] Compston A, Coles A. Multiple sclerosis. Lancet. 2008 Oct 25;372(9648):1502-17. doi: 10.1016/S0140-6736(08)61620-7. PMID 18970977
- [Background] ElSankari S, Baledent O, van Pesch V, Sindic C, de Broqueville Q, Duprez T. Concomitant analysis of arterial, venous, and CSF flows using phase-contrast MRI: a quantitative comparison between MS patients and healthy controls. J Cereb Blood Flow Metab. 2013 Sep;33(9):1314-21. doi: 10.1038/jcbfm.2013.95. Epub 2013 Jun 19. PMID 23778162